CLINICAL TRIAL: NCT06103032
Title: Long-term Survival of Breast-conserving Surgery Versus Mastectomy in Asymptomatic Screen-detected Unilateral and Bilateral, Unifocal and Multifocal, Young and Elderly Non-palpable Breast Cancer Among Chinese Women
Brief Title: Survival of BCS vs Mx in Asymptomatic Screen-detected NPBC
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-BSBM
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Segmental; Mastectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- a consecutive cohort of women with asymptomatic screen-detected non-palpable breast cancer: a consecutive cohort of women with asymptomatic screen-detected non-palpable breast cancer treated in Dept. Breast Surgery, PUMC Hospital from January 2003 to December 2017
  Interventions: Procedure: Breast Conserving Surgery; Procedure: Mastectomy

INTERVENTIONS:
Procedure: Breast Conserving Surgery — Patients undergoing breast conserving surgery
Procedure: Mastectomy — Patients undergoing mastectomy

SUMMARY:
We performed this study on a consecutive cohort of women with asymptomatic screen-detected NPBC. The clinicopathological characteristics, 10-year relapse-free survival (RFS) and overall survival (OS) were compared between BCS and Mx patients among different subgroups.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent must be obtained and documented according to the local regulatory requirements prior to beginning specific protocol procedures.

Age of at least 18 and at most 90 years. Performance status (Karnofsky-Index) >80%. Chemotherapy is necessary before or after surgery. No clinical evidence of local recurrence or distant metastases. Complete staging work-up within 3 months prior to registration. All patients must have (bilateral) mammography or breast MRI, chest X-ray; other tests may be performed as clinically indicated.

Life expectancy of at least 2 years, disregarding the diagnosis of cancer. Adequate organ function including normal red and white blood count, platelets, serum creatinine, bilirubin, and transaminases within normal range of the institution.

Patients must be available for and compliant to treatment and follow-up. Patients registered on this trial must be treated and followed up at the participating center.

Exclusion Criteria:

Known hypersensitivity reaction to the investigational compounds or incorporated substances.

Local recurrence and/or metastasis of breast cancer. No need of chemotherapy. Pregnant or lactating patients. Patients of childbearing potential must have a negative pregnancy test (urine or serum) within 14 days prior to registration.

Prior or concomitant secondary malignancy (except non-melanomatous skin cancer or carcinoma in situ of the uterine cervix) Any other serious medical pathology, such as congestive heart failure; unstable angina; history of myocardial infarction during the previous year; uncontrolled high risk arrhythmias Other serious illness or medical condition that may interfere with the understanding and giving of informed consent and the conduct of the study.

Concurrent treatment with other experimental drugs or any other anti-cancer therapy.

Males.

Ages: 18 Years to 90 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: a consecutive cohort of women with asymptomatic screen-detected non-palpable breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 1020 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
The clinicopathological characteristics were compared between BCS and Mx patients | 15 years
The prognosis was compared between BCS and Mx patients | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Qiang SUN, Dr., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
No sharing according to the privacy of patients.